CLINICAL TRIAL: NCT04323930
Title: Randomized Control Trial of the eyeWatch System as a First-Line Surgical Treatment of Glaucoma vs. MMC-Trabeculectomy
Brief Title: eyeWatch vs. Trabeculectomy RCT (evT)
Acronym: evT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr. Kaweh Mansouri (Other)
Collaborators: Manchester Royal Eye Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr. Kaweh Mansouri, MD MPH, Swiss Vision Network
Organization: Swiss Vision Network (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: evT-2020
Record Dates: First submitted 2020-03-20; First posted 2020-03-27 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Primary Glaucoma
MeSH Terms: interventions — Trabeculectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eyeWatch (Experimental)
  Interventions: Device: eyeWatch
- Trabeculectomy (Experimental)
  Interventions: Device: eyeWatch

INTERVENTIONS:
Device: eyeWatch — The eyeWatch system will be implanted as per the manufacturer's instruction, and trabeculectomy will be performed using mitomycin C as per standard surgical protocols.
  Other Names: Trabeculectomy

SUMMARY:
The confirm the performance and safety of the eyeWatch System as first-line filtering surgery and compare its outcomes to trabeculectomy

DETAILED DESCRIPTION:
Open-angle glaucoma is an ophthalmic disease often characterised by high intraocular pressures. Traditionally, glaucoma is treated using medication, however, more advanced or refractory glaucoma requires surgical treatment. In terms of surgery, the current gold-standard is trabeculectomy. Despite good efficacy, the technique carries relatively high rates of complications. The eyeWatch system has recently received CE-marking for the treatment of open-angle glaucoma. During its initial clinical trial, the eyeWatch system demonstrated good safety and efficacy profile. The present randomized control trial will assess its safety and efficacy against the current gold-standard: trabeculectomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 95 years,
* Diagnosis of primary open-angle glaucoma, pseudo-exfoliative glaucoma or pigmentary glaucoma in the study eye (based on [1] glaucomatous optic neuropathy and [2] visual field defects in keeping with optic disc appearance),
* Phakic or pseudophakic study eye,
* Indication for primary filtering surgery (defined as a corrected IOP ≥ 20 mmHg in the study eye, under maximally tolerated therapy on 2 consecutive measurements made on different days prior to surgery),
* Undergoing surgery and post-operative follow-up at one of the investigations centres: Montchoisi Clinic, Swiss Visio, Lausanne, Switzerland OR Manchester Royal Eye Hospital, Manchester, United-Kingdom,
* Patient agreed to sign the written inform consent prior to entering the study,
* Patient is able and willing to complete post-operative follow-up requirements.

Exclusion Criteria:

* Diagnosis of secondary glaucoma except for pseudo-exfoliative or pigmentary glaucoma (neovascular glaucoma, congenital glaucoma, uveitic glaucoma…),
* Previous filtering or tube surgery in the same eye (including trabeculectomy, deep-sclerectomy and all GDDs / excluding XEN gel stents, angle surgery, cataract surgery and all MIGS),
* Recent ophthalmic surgery (less than 3 months prior to inclusion) or indication for a combined procedure (no combined surgeries will be performed),
* Narrow iridocorneal angles defined as a Shaffer grade ≤ 2 or presence of iris bombé,
* Endothelial cell density < 1500 cells/mm²,
* Presence of other significant pathologies in the study eye (including extensive conjunctival thinning or scarring, optic neuropathy of non-glaucomatous etiology, retinal vein occlusion, retinal artery occlusion, corneal opacification or irregularities, ocular malformations such as microphthalmia, concurrent inflammation/infection),
* Proliferative or severe non-proliferative retinopathy in either eye,
* Any sign of past or present uveitis,
* Severe systemic disease or disabling conditions (including chronic renal failure, history of organ transplantation),
* Current or recent participation in another clinical trial (less than 3 months prior to inclusion),
* Pregnancy or breast-feeding,
* Inability to give informed consent to participate to a clinical investigation.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (mmHg) | pre-op to month 12
  The primary endpoint will be the change in intraocular pressure (mmHg) from pre-operative baseline to 12-month post-operatively. Intraocular pressure will be measure at each visit using Goldmann tonometry. Baseline intraocular pressure will be defined as the mean of the last two pre-operative measurements.
number of anti glaucoma medications | pre-op to month 12
  The number of anti-glaucoma medications will be reported for each visit and compared to the baseline.

SECONDARY OUTCOMES:
Visual acuity | baseline to month 12
  Visual acuity will be measured at each visit and compared to the baseline measurement.
visual field mean deviation | baseline to month 12
  Visual field mean deviation will be measured at each visit and compared to the baseline measurement.
endothelial cell density | baseline to month 12
  the number of endothelial cells will be measured at each visit and compared to the baseline measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- SwissVisio Montchoisi, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No